CLINICAL TRIAL: NCT07273799
Title: Comparison of Outcomes Between Topical Minoxidil Versus Oral Minoxidil for the Treatment of Androgenetic Alopecia
Acronym: mina
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Sohaib Ashraf, Consultant Cardiologist, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-TERC/NHRC-SZH/Int-SC/651
Record Dates: First submitted 2025-11-16; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Androgenic Alopecia
Keywords: Androgenic Alopecia; Minoxidil
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Disease Control (Placebo Comparator): Placebo spray and palcebo tablet
  Interventions: Drug: Placebo Spray; Drug: Placebo Tablet or Capsule
- Minoxidil Spray Arm (Active Comparator): Placebo tablet Mixidil spray
  Interventions: Drug: Minoxidil 5 % Topical Spray; Drug: Placebo Tablet or Capsule
- Minoxidil Tablet Arm (Active Comparator): Mixidil tablet placebo spray
  Interventions: Drug: minoxidil; Drug: Placebo Spray
- Minoxidil Tablet + Spray Arm (Experimental): Minoxidil spray Minoxidil Tablet
  Interventions: Drug: Minoxidil 5 % Topical Spray; Drug: minoxidil

INTERVENTIONS:
Drug: Minoxidil 5 % Topical Spray — Topical spray on hairs
  Arms: Minoxidil Spray Arm; Minoxidil Tablet + Spray Arm
Drug: minoxidil — Oral minoxidil 2.5mg
  Arms: Minoxidil Tablet + Spray Arm; Minoxidil Tablet Arm
Drug: Placebo Spray — placebo spray
  Arms: Disease Control; Minoxidil Tablet Arm
Drug: Placebo Tablet or Capsule — Placebo tablet
  Arms: Disease Control; Minoxidil Spray Arm

SUMMARY:
To compare the outcome of topical minoxidil 5% spray versus oral minoxidil 2.5 mg tablet for the treatment of androgenetic alopecia in males and females. Outcomes include efficacy of the treatment, measured by reduction in hair shedding, improvement in hair density and new hair growth as assessed by physican and patient assessment as well as safety, defined as incidence and severity of adverse events over a treatment period of 6 months

DETAILED DESCRIPTION:
This cohort, adaptive, randomized, double armed group, controlled, investigator-initiated interventional study is designed to demonstrate the superiority of a combination of Topical minoxidil vs oral minoxidil in patients suffering from androgenetic alopecia who consent to randomization following a new diagnosis in Pakistan.

Conditions Androgenetic Alopecia

Intervention/Treatment:

Drug: Oral Minoxidil Drug: Topical Minoxidil

ELIGIBILITY:
Inclusion Criteria:

* Patients with androgenic alopecia Norwood-Hamilton class 2-6 in males and Sinclair class 2-5 in females
* History of androgentic alopecia for at least 1 year
* 18 to 50 years of age
* Willing to provide informed consent
* Willing to not use any other hair loss treatment during the treatment period

Exclusion Criteria:

* History of cardiovascular disease
* Use of some other hair restoration therapy in the past 6 months such as minoxidil, finasteride or PRP
* Presence of other causes of alopecia (e.g., alopecia areata, scarring alopecia).
* Pregnant and lactating females
* Previous Hair Transplantation
* Patients with a known hypersensitivity to the study drug or class of study drug
* Patients with co-morbid conditions like chronic liver disease, chronic kidney disease, neurological or psychiatric disorders
* Presence of any other autoimmune disease (especially thyroid disease)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of drug | 6 months
  The effectiveness of the treatment in terms of reduction in hair shedding, improvement in hair density, and new hair growth will be measured by a standardised seven point scale for physician photographic assessment and patient self assessment.
Physician Photographic Assessment Scale | 6 months
  (+3 = Excellent Improvement, +2 = moderately improvement , +1 = mild improvement, 0 = no change, -1 = mild worsening, -2 =moderate worsening, -3 = severe worsening)
Patient Satisfaction Scale | 6 months
  -3 Very Unsatisfied, -2 Moderately Unsatisfied, -1 Slightly Unsatisfied, 0 No Change, 1 Slightly Satisfied, 2 Moderately Satisfied, 3 Very Satisfied

SECONDARY OUTCOMES:
Drug Safety | 6 months
  It is defined as the incidence and severity of adverse events associated with oral and topical minoxidil over the treatment period. This includes localised adverse effects, such as eczema, scalp irritation, light headedness, headache or hypertrichosis, and systemic adverse effects, such as tachycardia, fluid retention and allergic reactions. All information will be recorded in a predesigned proforma.
Severity of adverse eﬀect (mild, moderate, severe) | 6 months
  Each adverse effect will be categorized as Mild, Moderate and Severe:
  Mild: No interference with daily activities; may include mild scalp itching or irritation Moderate: Requires intervention (e.g., symptomatic treatment) but allows continuation of minoxidil. Severe: Interferes significantly with daily activities or presents a risk to the patient's health, potentially requiring cessation of treatment (e.g. persistent tachycardia or severe allergic reaction).

IPD SHARING:
Plan to Share IPD: No